CLINICAL TRIAL: NCT04119310
Title: Lumbar Thrust-mobilization Effects on Hip Strength and Anterior Knee Pain, a Double Blind Randomized Control Trial
Brief Title: Lumbar Thrust-mobilization Effects on Hip Strength and Anterior Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Messiah College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BergmannHumphrey
Record Dates: First submitted 2019-10-01; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two interventions, thrust-mobilization or sham mobilization.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind: The subjects will not know what intervention they are receiving - same generic script is provided. One Investigator is performing all pre and post-tests without knowledge of intervention, the other investigator is opening the envelope and providing the intervention behind a screen without knowledge of test results. This investigator will record the subjects assigned # and which intervention they received. Investigators will record data on spreadsheet separately.
  The outcomes will be evaluated by a masked outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar thrust-mobilization (Experimental): The investigator will perform a lumbar thrust-mobilization with the subject in right and then left sidelying position
  Interventions: Other: Lumbar-thrust mobilization
- Sham-mobilization (Sham Comparator): No lumbar-thrust mobilization will be performed. Subject will receive simple passive inter-vertebral range of motion.
  Interventions: Other: Sham thrust-mobilization

INTERVENTIONS:
Other: Lumbar-thrust mobilization — The intervention group will receive passive spinal rotational grade V thrust-mobilization, based on Maitland's approach. The intervention will be performed with the subject in right sidelying and left sidelying. The operator's palpating hand is placed over the L2-3 intervertebral space, and the other hand bends both legs of the participant up to the range at which the L2-3 midposition is found. The participant is then asked to straighten the lower leg and hook the upper leg over it with the upper leg's knee positioned over the side of the plinth. While the lower component is kept still, the participant's trunk is rotated until the hip starts to lift off from the plinth. The bottom hand and uppermost hand rest under a pillow and the chest wall, respectively. With the starting position settled, the operator stands behind the participant, takes up the slack within the spine and then provides a grade V thrust- mobilization while stabilizing the uppermost shoulder.
  Other Names: Grade 5 mobilization, manipulation
  Arms: Lumbar thrust-mobilization
Other: Sham thrust-mobilization — Subjects are positioned in right sidelying. The experimenter holds both knees with one arm while placing their opposite hand on the participant's lumbar spine. The experimenter performs 1 min of ﬂexion and extension passive range of motion without reaching physiological end range in either direction of movement. This is repeated with the subject in left sidelying.
  Arms: Sham-mobilization

SUMMARY:
The purpose of this study is to investigate changes in lateral hip muscle strength as well as self-reported pain during the performance of three functional tests in patients with anterior knee pain following a lumbopelvic thrust-mobilization.

Hypothesis(es):

Lumbar thrust-mobilization will lead to increased lateral hip strength and decreased anterior knee pain during 3 functional activities (single leg step down, functional squat, drop jump).

DETAILED DESCRIPTION:
The participant will complete a medical history form and undergo a brief physical exam of the lumbar spine and knees to include: lumbar range of motion and mobility testing, knee range of motion, palpation, and knee mobility testing. The participant will complete a hip strength test utilizing the Biodex System 4 Pro®. The participant will then perform three activities (single leg step down, squat, and drop jump from a 2 foot platform) and provide a self-reported knee pain measure with each activity. A sealed envelope indicating the intervention to be received will be given to the participant. An investigator blinded to the pre and post-measures will open the envelope indicating the intervention to be performed. The participant will be blinded to which intervention group they are categorized to. Th e participant will be positioned on a high-low treatment table to receive the assigned intervention. The participant will be positioned to receive either intervention 1 (thrust mobilization) or 2 (sham mobilization). The participant will either receive the thrust-mobilization or sham mobilization up to 2 times on the left and right side. An immediate re-test of hip strength will be conducted followed by performing the same three functional activities (single leg step down, squat, and drop jump from a 2 foot platform) while providing a self-reported pain measure after each activity. Follow-up measures at 15 minutes post-intervention and the final measure at 30 minutes post-intervention will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between the ages of 18 and 25 with non-traumatic anterior knee pain
* Able read and write in English
* Clearly understand the informed consent form

Exclusion Criteria:

* Low back pain
* Pregnant or may be pregnant
* Previously diagnosed with spondylolisthesis,
* Previously diagnosed with a herniated disc,
* Signs and symptoms of nerve root compression
* History of spine surgery
* History of knee surgery
* History of cancer
* History of compression fracture
* History of osteoporosis
* History of osteopenia
* History of a systemic disease
* History of a connective tissue disease
* History of a neurological disease
* Pain with pre-manipulative hold
* Positive findings on medical history form, or physical exam
* Presence of anxiety during the procedure

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in lateral hip strength | Pre-intervention, immediately following intervention, 15 min post-intervention & 30 min post-intervention
  lateral isometric hip strength will be measured with Biodex system 4
Change in pain with single leg step down | Pre-intervention, immediately following intervention, 15 min post-intervention & 30 min post-intervention
  Subject will provide level of anterior knee pain via Visual Analogue Scale (VAS) while performing a single leg step down.
  The VAS pain scale is a 0 to 10 scale, 0 indicates no pain, 5 indicates distressing pain, 10 indicates unbearable pain. Any whole number between 0 and 10 may be chosen. 0 is better and 10 is worse.
Change in pain with double leg squat | Pre-intervention, immediately following intervention, 15 min post-intervention & 30 min post-intervention
  Subject will provide level of anterior knee pain via Visual Analogue Scale (VAS) while performing a double leg squat.
  The VAS pain scale is a 0 to 10 scale, 0 indicates no pain, 5 indicates distressing pain, 10 indicates unbearable pain. Any whole number between 0 and 10 may be chosen. 0 is better and 10 is worse.
Change in pain with drop jump from 2 foot platform | Pre-intervention, immediately following intervention, 15 min post-intervention & 30 min post-intervention
  Subject will provide level of anterior knee pain via Visual Analogue Scale (VAS) while performing a drop jump from a 2 foot platform.
  The VAS pain scale is a 0 to 10 scale, 0 indicates no pain, 5 indicates distressing pain, 10 indicates unbearable pain. Any whole number between 0 and 10 may be chosen. 0 is better and 10 is worse.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saltychev M, Dutton RA, Laimi K, Beaupre GS, Virolainen P, Fredericson M. Effectiveness of conservative treatment for patellofemoral pain syndrome: A systematic review and meta-analysis. J Rehabil Med. 2018 May 8;50(5):393-401. doi: 10.2340/16501977-2295. PMID 29392329
- [Background] Bizzini M, Childs JD, Piva SR, Delitto A. Systematic review of the quality of randomized controlled trials for patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2003 Jan;33(1):4-20. doi: 10.2519/jospt.2003.33.1.4. PMID 12570282
- [Background] Powers CM. The influence of abnormal hip mechanics on knee injury: a biomechanical perspective. J Orthop Sports Phys Ther. 2010 Feb;40(2):42-51. doi: 10.2519/jospt.2010.3337. PMID 20118526
- [Background] Iverson CA, Sutlive TG, Crowell MS, Morrell RL, Perkins MW, Garber MB, Moore JH, Wainner RS. Lumbopelvic manipulation for the treatment of patients with patellofemoral pain syndrome: development of a clinical prediction rule. J Orthop Sports Phys Ther. 2008 Jun;38(6):297-309; discussion 309-12. doi: 10.2519/jospt.2008.2669. Epub 2008 Jan 22. PMID 18515959
- [Background] Sutlive TG, Mitchell SD, Maxfield SN, McLean CL, Neumann JC, Swiecki CR, Hall RC, Bare AC, Flynn TW. Identification of individuals with patellofemoral pain whose symptoms improved after a combined program of foot orthosis use and modified activity: a preliminary investigation. Phys Ther. 2004 Jan;84(1):49-61. PMID 14992676
- [Background] Boling M, Padua D, Marshall S, Guskiewicz K, Pyne S, Beutler A. Gender differences in the incidence and prevalence of patellofemoral pain syndrome. Scand J Med Sci Sports. 2010 Oct;20(5):725-30. doi: 10.1111/j.1600-0838.2009.00996.x. PMID 19765240
- [Background] Lesher JD, Sutlive TG, Miller GA, Chine NJ, Garber MB, Wainner RS. Development of a clinical prediction rule for classifying patients with patellofemoral pain syndrome who respond to patellar taping. J Orthop Sports Phys Ther. 2006 Nov;36(11):854-66. doi: 10.2519/jospt.2006.2208. PMID 17154139
- [Background] Robinson RL, Nee RJ. Analysis of hip strength in females seeking physical therapy treatment for unilateral patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2007 May;37(5):232-8. doi: 10.2519/jospt.2007.2439. PMID 17549951
- [Background] Cowan SM, Hodges PW, Bennell KL, Crossley KM. Altered vastii recruitment when people with patellofemoral pain syndrome complete a postural task. Arch Phys Med Rehabil. 2002 Jul;83(7):989-95. doi: 10.1053/apmr.2002.33234. PMID 12098160
- [Background] McCarthy MM, Strickland SM. Patellofemoral pain: an update on diagnostic and treatment options. Curr Rev Musculoskelet Med. 2013 Jun;6(2):188-94. doi: 10.1007/s12178-013-9159-x. PMID 23456237
- [Background] Dixit S, DiFiori JP, Burton M, Mines B. Management of patellofemoral pain syndrome. Am Fam Physician. 2007 Jan 15;75(2):194-202. PMID 17263214
- [Background] Pappas E, Wong-Tom WM. Prospective Predictors of Patellofemoral Pain Syndrome: A Systematic Review With Meta-analysis. Sports Health. 2012 Mar;4(2):115-20. doi: 10.1177/1941738111432097. PMID 23016077
- [Background] Waryasz GR, McDermott AY. Patellofemoral pain syndrome (PFPS): a systematic review of anatomy and potential risk factors. Dyn Med. 2008 Jun 26;7:9. doi: 10.1186/1476-5918-7-9. PMID 18582383
- [Background] Witvrouw E, Lysens R, Bellemans J, Cambier D, Vanderstraeten G. Intrinsic risk factors for the development of anterior knee pain in an athletic population. A two-year prospective study. Am J Sports Med. 2000 Jul-Aug;28(4):480-9. doi: 10.1177/03635465000280040701. PMID 10921638
- [Background] Powers CM. Rehabilitation of patellofemoral joint disorders: a critical review. J Orthop Sports Phys Ther. 1998 Nov;28(5):345-54. doi: 10.2519/jospt.1998.28.5.345. PMID 9809282
- [Background] Crossley K, Bennell K, Green S, McConnell J. A systematic review of physical interventions for patellofemoral pain syndrome. Clin J Sport Med. 2001 Apr;11(2):103-10. doi: 10.1097/00042752-200104000-00007. PMID 11403109
- [Background] Lake DA, Wofford NH. Effect of therapeutic modalities on patients with patellofemoral pain syndrome: a systematic review. Sports Health. 2011 Mar;3(2):182-9. doi: 10.1177/1941738111398583. PMID 23016007
- [Background] Crossley K, Bennell K, Green S, Cowan S, McConnell J. Physical therapy for patellofemoral pain: a randomized, double-blinded, placebo-controlled trial. Am J Sports Med. 2002 Nov-Dec;30(6):857-65. doi: 10.1177/03635465020300061701. PMID 12435653
- [Background] Tyler TF, Nicholas SJ, Mullaney MJ, McHugh MP. The role of hip muscle function in the treatment of patellofemoral pain syndrome. Am J Sports Med. 2006 Apr;34(4):630-6. doi: 10.1177/0363546505281808. Epub 2005 Dec 19. PMID 16365375
- [Background] Lowry CD, Cleland JA, Dyke K. Management of patients with patellofemoral pain syndrome using a multimodal approach: a case series. J Orthop Sports Phys Ther. 2008 Nov;38(11):691-702. doi: 10.2519/jospt.2008.2690. PMID 18978450
- [Background] Mascal CL, Landel R, Powers C. Management of patellofemoral pain targeting hip, pelvis, and trunk muscle function: 2 case reports. J Orthop Sports Phys Ther. 2003 Nov;33(11):647-60. doi: 10.2519/jospt.2003.33.11.647. PMID 14669960
- [Background] Fukuda TY, Rossetto FM, Magalhaes E, Bryk FF, Lucareli PR, de Almeida Aparecida Carvalho N. Short-term effects of hip abductors and lateral rotators strengthening in females with patellofemoral pain syndrome: a randomized controlled clinical trial. J Orthop Sports Phys Ther. 2010 Nov;40(11):736-42. doi: 10.2519/jospt.2010.3246. PMID 21041965
- [Background] Pickar JG. Neurophysiological effects of spinal manipulation. Spine J. 2002 Sep-Oct;2(5):357-71. doi: 10.1016/s1529-9430(02)00400-x. PMID 14589467
- [Background] Espi-Lopez GV, Arnal-Gomez A, Balasch-Bernat M, Ingles M. Effectiveness of Manual Therapy Combined With Physical Therapy in Treatment of Patellofemoral Pain Syndrome: Systematic Review. J Chiropr Med. 2017 Jun;16(2):139-146. doi: 10.1016/j.jcm.2016.10.003. Epub 2016 Nov 22. PMID 28559754
- [Background] Grindstaff TL, Hertel J, Beazell JR, Magrum EM, Kerrigan DC, Fan X, Ingersoll CD. Lumbopelvic joint manipulation and quadriceps activation of people with patellofemoral pain syndrome. J Athl Train. 2012 Jan-Feb;47(1):24-31. doi: 10.4085/1062-6050-47.1.24. PMID 22488227
- [Background] Grindstaff TL, Hertel J, Beazell JR, Magrum EM, Ingersoll CD. Effects of lumbopelvic joint manipulation on quadriceps activation and strength in healthy individuals. Man Ther. 2009 Aug;14(4):415-20. doi: 10.1016/j.math.2008.06.005. Epub 2008 Sep 20. PMID 18805726
- [Background] Sanders GD, Nitz AJ, Abel MG, Symons TB, Shapiro R, Black WS, Yates JW. Effects of Lumbosacral Manipulation on Isokinetic Strength of the Knee Extensors and Flexors in Healthy Subjects: A Randomized, Controlled, Single-Blind Crossover Trial. J Chiropr Med. 2015 Dec;14(4):240-8. doi: 10.1016/j.jcm.2015.08.002. Epub 2015 Nov 6. PMID 26793035
- [Background] Yuen TS, Lam PY, Lau MY, Siu WL, Yu KM, Lo CN, Ng J. Changes in Lower Limb Strength and Function Following Lumbar Spinal Mobilization. J Manipulative Physiol Ther. 2017 Oct;40(8):587-596. doi: 10.1016/j.jmpt.2017.07.003. PMID 29187310
- [Background] Hillermann B, Gomes AN, Korporaal C, Jackson D. A pilot study comparing the effects of spinal manipulative therapy with those of extra-spinal manipulative therapy on quadriceps muscle strength. J Manipulative Physiol Ther. 2006 Feb;29(2):145-9. doi: 10.1016/j.jmpt.2005.12.003. PMID 16461174
- [Background] Suter E, McMorland G, Herzog W, Bray R. Conservative lower back treatment reduces inhibition in knee-extensor muscles: a randomized controlled trial. J Manipulative Physiol Ther. 2000 Feb;23(2):76-80. PMID 10714531
- [Background] Suter E, McMorland G, Herzog W, Bray R. Decrease in quadriceps inhibition after sacroiliac joint manipulation in patients with anterior knee pain. J Manipulative Physiol Ther. 1999 Mar-Apr;22(3):149-53. doi: 10.1016/S0161-4754(99)70128-4. PMID 10220713